CLINICAL TRIAL: NCT02646462
Title: Systematic Lymph Node Sampling and Analysis in Patients Undergoing Radical Resection for Pancreatic Cancer. A National Danish Study
Brief Title: Systematic Lymph Node Sampling and Analysis in Patients With Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Michael Bau Mortensen (Other)
Responsible Party: Sponsor-Investigator, Michael Bau Mortensen, professor, MD, PhD, DMSci, Odense University Hospital
Organization: Odense University Hospital (Other)
Other Study IDs: 24
Record Dates: First submitted 2015-06-05; First posted 2016-01-05 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Pancreatic Cancer
Keywords: pancreas adenocarcinoma, lymph node metastases
MeSH Terms: conditions — Pancreatic Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Prospective investigation of the ratio between malignant and total number of lymph nodes in predefined lymph node stations in patients resected for pancreatic adenocarcinoma. A national Danish project.

DETAILED DESCRIPTION:
Lymph nodes will be sampled from the following stations in patients with adenocarcinomas of the pancreas Group 6: Infrapyloric lymph nodes (IP) Group 8: Lymph nodes around the common hepatic artery (CHA) Group 12: Lymph nodes of the hepatoduodenal ligament (HDL) Group 13: Posterior pancreaticoduodenal lymph nodes Group 14: Lymph nodes around the superior mesenteric artery (SMA) Group 17: Anterior pancreaticoduodenal lymph nodes

ELIGIBILITY:
Inclusion Criteria:

Bioptic verified pancreatic adenocarcinoma or periampullary adenocarcinoma (within 20mm of the papilla)

Exclusion Criteria:

Patients with non-adenocarcinoma tumors of the pancreas or periampullary region

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bioptic verified pancreatic adenocarcinoma or periampullary adenocarcinoma (within 20mm of the papilla) referred for pancreas resection
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Ratio of malignant/total number of lymph nodes | 12 months
  Ratio between malignant and total number of lymph nodes in predefined lymph node stations

SECONDARY OUTCOMES:
Number of N1 patients | 12 months
  Number of patients with malignant lymph nodes in predefined lymph node stations

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: No